CLINICAL TRIAL: NCT02960373
Title: Dried Fruit as a Means for Lowering the Glycemic Response to High Glycemic Index-carbohydrate Foods
Brief Title: Dried Fruit and Postprandial Glycemia Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: International Nut and Dried Fruit Council (INC) (Unknown); The National Dried Fruit Trade Association (NDFTA) (Unknown); Glycemia Consulting Inc. (Unknown)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, Staff Physician, Scientist, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: INC-Dried Fruit Trial 2016
Record Dates: First submitted 2016-11-01; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: PreDiabetes; Diabetes Mellitus; Dysglycemia
Keywords: Dried fruit; Glycemic Index; Catalytic dose; Glycemic response; Fructose; Postprandial; Randomized clinical trial; Carbohydrate metabolism
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- White Bread (Control) (Active Comparator): Participants will consume a test meal containing white bread (dose: 50g available carbohydrate) at three study visits.
  Interventions: Other: White Bread (Control)
- Dried Fruit - Glycemic Index (Experimental): Participants will consume a test meal containing one variety of dried fruit (dose: 50g available carbohydrate) per visit for four visits. Varieties include raisins, sultanas, dates, and apricots.
  Interventions: Other: Dried Fruit - Glycemic Index
- Catalytic Fructose Dose Effect (Experimental): Participants will consume a test meal containing white bread (dose: 50g available carbohydrate) and one variety of dried fruit (dose: 7g fructose) per visit for four visits. Varieties of dried fruit include: raisins, sultanas, dates, and apricots.
  Interventions: Other: Catalytic Fructose Dose Effect
- High GI Displacement Effect (Experimental): Participants will consume a test meal containing white bread (dose: 25g available carbohydrate) and one variety of dried fruit (dose: 25g available carbohydrate) per visit for four visits. Varieties of dried fruit include: raisins, sultanas, dates, and apricots.
  Interventions: Other: High GI Displacement Effect

INTERVENTIONS:
Other: White Bread (Control) — A randomized multiple-crossover acute-feeding trial design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 day washout period.
  Arms: White Bread (Control)
Other: Dried Fruit - Glycemic Index — A randomized multiple-crossover acute-feeding trial design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 day washout period.
  Arms: Dried Fruit - Glycemic Index
Other: Catalytic Fructose Dose Effect — A randomized multiple-crossover acute-feeding trial design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 day washout period.
  Arms: Catalytic Fructose Dose Effect
Other: High GI Displacement Effect — A randomized multiple-crossover acute-feeding trial design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 day washout period.
  Arms: High GI Displacement Effect

SUMMARY:
Dried fruits show promising potential for the management of blood glucose. Previous trials have reported beneficial effects of raisins on post-prandial glucose and insulin responses in healthy individuals when compared with white bread. However, to date there is limited data evaluating the potential beneficial effects of other dried fruits (i.e. sultanas, dates and apricots). It is also unclear whether dried fruits can be used to lower the postprandial glycemic responses to high-GI carbohydrate foods by either displacing available carbohydrate (displacement effect) or providing 'catalytic' doses of fructose ('catalytic' fructose effect). To address these questions, the investigators propose to assess the GI of 4 common types of dried fruit (raisins, sultanas, dates, apricots) (GI effect) and their ability to decrease the postprandial glycemic response to white bread by either partially displacing available carbohydrate (displacement effect) or by providing a 'catalytic' dose of fructose ('catalytic' fructose effect).

DETAILED DESCRIPTION:
BACKGROUND:

All studies assessing the glycemic index (GI) of traditional dried fruit show that they are low-to-moderate GI foods and that the insulin response is proportional to their GI. A recent study compared the glycemic response of two doses of raisins (28 and 69g) versus white bread showing that both doses of raisins significantly reduced post-prandial glucose and insulin levels compared with white bread. However, the effect of combining dried fruits with high-GI carbohydrate foods has never been addressed. The potential impact of combining nuts (i.e. pistachios) and high-GI carbohydrate foods has already analyzed with positive results. The investigators found that a dose of 56g of pistachios consumed alone had a minimal effect on post-prandial glycemia, but when taken with a high-carbohydrate meal attenuated the relative glycemic response. Although foods with high fibre content generally have a low-GI, other factors also contribute to a food's glycemic response. Factors thought to contribute to the glycemic response of dried fruits include the viscous texture when chewed; their whole food matrix; the presence of phenolic compounds and organic acids and the type of sugar present. In the case of dried fruit, about 50% fructose (low-GI) is present. Therefore, the consumption of dried fruit with high-carbohydrate foods may lead to glycemic control benefits by lowering the GI of a food. In addition to potentially lowering the GI of a food, dried fruits may also affect glycemic control by providing 'catalytic' doses of fructose. Fructose, through its metabolite fructose-1-P, has been shown to have "catalytic" effects on hepatic glucose metabolism by inducing glucokinase activity in hepatocytes. In specific, fructose-1-P displaces fructose-6-P from glucokinase's regulatory binding protein in the nucleus causing the release of glucokinase from its regulatory protein, allowing it to translocate to the cytosol, resulting in increased phosphorylation of glucose. Infusion studies in humans have shown that this mechanism relates to a ~30% decrease in hepatic glucose output under hyperglycemic conditions in participants with type 2 diabetes (T2D) and a ~3-fold increase in glycogen synthesis by C13-nuclear magnetic resonance (NMR) spectroscopy under euglycemic conditions in healthy people. Clinical translation of these findings has proven promising. Catalytic doses of fructose at 7.5g and 10g have been shown to decrease the postprandial glycemic responses to high GI meals (oral glucose, maltodextrins, or mashed potatoes) from ~15-30% in healthy participants and those with pre-diabetes or diabetes . These acute effects have been shown to be sustainable over the longer term as well. Systematic reviews and meta-analyses of controlled feeding trials have shown that small doses of fructose in exchange for other carbohydrates decreases HbA1c at a level which exceeds the clinically meaningful threshold of 0.3% proposed by the Federal Drug Administration (FDA) for the development of new oral anti-hyperglycemic agents. Therefore, the consumption of dried fruit with high-carbohydrate foods may lead to glycemic control benefits by acting as a vehicle for 'catalytic' doses of fructose.

OBJECTIVES:

To investigate the effect of using dried fruit to modify the glycemic response of high GI foods, the investigators propose the following 3 objectives:

1. To assess the GI of 4 common types of dried fruit (raisins, sultanas, dates, apricots) (GI effect)
2. To assess the ability of the 4 common types of dried fruit (raisins, sultanas, dates, apricots) to decrease the postprandial glycemic response to white bread by displacing half of the available carbohydrate (displacement effect)
3. To assess the ability of the 4 common types of dried fruit (raisins, sultanas, dates, apricots) to decrease the postprandial glycemic response to white bread by providing a 'catalytic' dose (7.5g) of fructose ('catalytic' fructose effect)

PARTICIPANTS:

The investigators will include male or non-pregnant female participants aged 18-75 years and who are otherwise healthy.

DESIGN:

The trial will use a randomized multiple crossover acute-feeding design in which each participants acts as their own control.

PROTOCOL:

The protocol will follow ISO 26642:2010(en), "Food products - Determination of the glycaemic index (GI) and recommendation for food classification". All participants will complete all test and control foods in the study series. An individual participant will normally complete 1 to 3 tests per week with at least one day in between. Participants will be studied between 7:00 and 9:30am after an overnight fast of 10-14h. On each test occasion the subject will be weighed, and two fasting blood samples will be obtained at -5 minute (min) intervals by finger-prick. Then the subject will start to consume a test meal. At the first bite a timer will be started and additional blood samples will be taken at 15, 30, 45, 60, 90 and 120 min after the start of the meal. Before and during the test, a blood glucose test record will be filled out with the subject's initials, ID number, date, body weight, test meal, time they start to eat, time it took to eat, time and composition of last meal, and any unusual activities. During the 2 hours the test subjects will remain seated.

BLOOD SAMPLES:

Each finger-prick sample consists of a total of 2-3 drops of blood obtained by finger prick and will be divided into two separate vials. The 2 to 3 drops of capillary blood will be collected into flat-bottomed 5ml plastic tubes with a push cap containing a small amount of sodium fluoride and potassium oxalate as an anticoagulant and preservative. These samples will be used for analyzing capillary blood glucose levels. The finger-prick samples for glucose analysis will initially be placed in the refrigerator and at the end of two hours, placed in a -20°C freezer until analysis which will be performed within a week. Glucose analysis will be done using a YSI model 2300 STAT analyzer (Yellow Springs, OH). Each subject will participate in a total of 15 separate test meals: 3 white bread control meals and 3 dried fruit treatments (dried fruit - GI effect, dried fruit -displacement effect, and dried fruit - 'catalytic' fructose effect) for each of the 4 dried fruits (raisins, sultanas, dates and apricots) (Figure 1). The order of the test meals will be randomized by a coordinator blinded to the treatment allocation. Test meals will be separated by a minimum of a 1-day washout.

STATISTICAL ANALYSES:

Blood glucose areas will be calculated as the incremental area under the curve (iAUC) using the trapezoidal rule with peak heights as maximal incremental rises in glucose. The glycemic indices of the test meals will be calculated using the 3 bread meals as the reference food. Pairwise differences in GI between the white bread control and the 3 dried fruit treatments (dried fruit - GI effect, dried fruit - GI displacement effect, and dried fruit - 'catalytic' fructose effect) for each of the 4 dried fruits (raisins, sultanas, dates and apricots) will be assessed by the Dunnett's test in SAS (SAS Inst. Version 8.2; Gary, NC).

EXPECTED RESULTS:

The investigators expect that dried fruit will have a low-to-moderate GI and will reduce postprandial glycemic responses when consumed in combination with high-GI foods in comparison to high-GI foods alone. The specific aims of our study are: (1) to quantify the GI of 4 different types of dried fruit (raisins, sultanas, dates, apricots) (GI effect); and (2) to assess the ability of these 4 dried fruits to decrease the postprandial glycemic response to white bread by either partially displacing available carbohydrate (displacement effect); or (3) by providing a 'catalytic' dose of fructose ('catalytic' fructose effect). The proposed study will help to identify mechanisms by which dried fruits can improve postprandial glycemia when consumed in combination with high-GI carbohydrate foods by assessing a glucose displacement mechanism along with a 'catalytic' fructose mechanism. The results will stimulate important industry innovation and improve the design of future clinical investigations that will ultimately lead to the use of dried fruits as an effective tool to modify the glycemic response of high carbohydrate foods and with it longer-term glycemic control in people with or at risk for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and/or non-pregnant females aged 18-75 years and in good health

Exclusion Criteria:

* Age less than 18 years or greater than 75 years
* BMI<18.5kg/m2 or >30kg/m2
* Known history of HIV, liver disease, kidney disease, thyroid disease, diabetes, heart disease or or any other major illnesses that may affect carbohydrate metabolism
* Subjects using medications which might, either: 1) make participation dangerous to the subject or to others, or 2) affect the results
* Subjects who cannot or will not comply with the experimental procedures or do not follow the clinic's safety guidelines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic index (GI) | Up to 120min

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD PhD FRCPC, Principal Investigator — University of Toronto, St. Michael's Hospital; Cyril Kendall, PhD, Principal Investigator — University of Toronto
Locations (1):
- GI Labs, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esfahani A, Lam J, Kendall CW. Acute effects of raisin consumption on glucose and insulin reponses in healthy individuals. J Nutr Sci. 2014 Jan 7;3:e1. doi: 10.1017/jns.2013.33. eCollection 2014. PMID 25191601
- [Background] University of Sydney, Online Glycemic Index Database. Accessed December 02 2015. URL Www.glycemicindex.com n.d.
- [Background] Kendall CW, Josse AR, Esfahani A, Jenkins DJ. The impact of pistachio intake alone or in combination with high-carbohydrate foods on post-prandial glycemia. Eur J Clin Nutr. 2011 Jun;65(6):696-702. doi: 10.1038/ejcn.2011.12. Epub 2011 Mar 2. PMID 21364607
- [Background] Kim Y, Hertzler SR, Byrne HK, Mattern CO. Raisins are a low to moderate glycemic index food with a correspondingly low insulin index. Nutr Res. 2008 May;28(5):304-8. doi: 10.1016/j.nutres.2008.02.015. PMID 19083424
- [Background] Agius L, Peak M. Intracellular binding of glucokinase in hepatocytes and translocation by glucose, fructose and insulin. Biochem J. 1993 Dec 15;296 ( Pt 3)(Pt 3):785-96. doi: 10.1042/bj2960785. PMID 8280078
- [Background] Van Schaftingen E, Detheux M, Veiga da Cunha M. Short-term control of glucokinase activity: role of a regulatory protein. FASEB J. 1994 Apr 1;8(6):414-9. doi: 10.1096/fasebj.8.6.8168691.
- [Background] Detheux M, Vandercammen A, Van Schaftingen E. Effectors of the regulatory protein acting on liver glucokinase: a kinetic investigation. Eur J Biochem. 1991 Sep 1;200(2):553-61. doi: 10.1111/j.1432-1033.1991.tb16218.x. PMID 1889418
- [Background] Vandercammen A, Detheux M, Van Schaftingen E. Binding of sorbitol 6-phosphate and of fructose 1-phosphate to the regulatory protein of liver glucokinase. Biochem J. 1992 Aug 15;286 ( Pt 1)(Pt 1):253-6. doi: 10.1042/bj2860253. PMID 1520277
- [Background] Hawkins M, Gabriely I, Wozniak R, Vilcu C, Shamoon H, Rossetti L. Fructose improves the ability of hyperglycemia per se to regulate glucose production in type 2 diabetes. Diabetes. 2002 Mar;51(3):606-14. doi: 10.2337/diabetes.51.3.606. PMID 11872657
- [Background] Petersen KF, Laurent D, Yu C, Cline GW, Shulman GI. Stimulating effects of low-dose fructose on insulin-stimulated hepatic glycogen synthesis in humans. Diabetes. 2001 Jun;50(6):1263-8. doi: 10.2337/diabetes.50.6.1263. PMID 11375325
- [Background] Moore MC, Cherrington AD, Mann SL, Davis SN. Acute fructose administration decreases the glycemic response to an oral glucose tolerance test in normal adults. J Clin Endocrinol Metab. 2000 Dec;85(12):4515-9. doi: 10.1210/jcem.85.12.7053. PMID 11134101
- [Background] Heacock PM, Hertzler SR, Wolf BW. Fructose prefeeding reduces the glycemic response to a high-glycemic index, starchy food in humans. J Nutr. 2002 Sep;132(9):2601-4. doi: 10.1093/jn/132.9.2601. PMID 12221216
- [Background] Iida T, Kishimoto Y, Yoshikawa Y, Hayashi N, Okuma K, Tohi M, Yagi K, Matsuo T, Izumori K. Acute D-psicose administration decreases the glycemic responses to an oral maltodextrin tolerance test in normal adults. J Nutr Sci Vitaminol (Tokyo). 2008 Dec;54(6):511-4. doi: 10.3177/jnsv.54.511. PMID 19155592
- [Background] Hayashi N, Iida T, Yamada T, Okuma K, Takehara I, Yamamoto T, Yamada K, Tokuda M. Study on the postprandial blood glucose suppression effect of D-psicose in borderline diabetes and the safety of long-term ingestion by normal human subjects. Biosci Biotechnol Biochem. 2010;74(3):510-9. doi: 10.1271/bbb.90707. Epub 2010 Mar 7. PMID 20208358
- [Background] Moore MC, Davis SN, Mann SL, Cherrington AD. Acute fructose administration improves oral glucose tolerance in adults with type 2 diabetes. Diabetes Care. 2001 Nov;24(11):1882-7. doi: 10.2337/diacare.24.11.1882. PMID 11679451
- [Background] Sievenpiper JL, Chiavaroli L, de Souza RJ, Mirrahimi A, Cozma AI, Ha V, Wang DD, Yu ME, Carleton AJ, Beyene J, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. 'Catalytic' doses of fructose may benefit glycaemic control without harming cardiometabolic risk factors: a small meta-analysis of randomised controlled feeding trials. Br J Nutr. 2012 Aug;108(3):418-23. doi: 10.1017/S000711451200013X. Epub 2012 Feb 21. PMID 22354959
- [Background] Cozma AI, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Wang DD, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on glycemic control in diabetes: a systematic review and meta-analysis of controlled feeding trials. Diabetes Care. 2012 Jul;35(7):1611-20. doi: 10.2337/dc12-0073. PMID 22723585
- [Background] Guidance for Industry Diabetes Mellitus: Developing Drugs and Therapeutic Biologics for Treatment and Prevention (DRAFT GUIDANCE), U.S Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Editor. 2008: Rockville, MD. p. 1-30.
- [Derived] Viguiliouk E, Jenkins AL, Blanco Mejia S, Sievenpiper JL, Kendall CWC. Effect of dried fruit on postprandial glycemia: a randomized acute-feeding trial. Nutr Diabetes. 2018 Dec 11;8(1):59. doi: 10.1038/s41387-018-0066-5. PMID 30531821